CLINICAL TRIAL: NCT04762472
Title: The Impact of Particulate Matters Air Pollution on Accelerated Atherosclerosis: A Montelukast Interventional Study for Atherosclerosis Prevention in Modernizing China
Brief Title: Air Pollution (PM2.5) on Accelerated Atherosclerosis: A Montelukast Interventional Study in Modernizing China
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: People's Hospital of Chongqing (Other); Hong Kong University of Science and Technology (Other); Chongqing Medical University (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Kam Sang WOO, Adjunct Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-398
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Atherosclerosis, Coronary
Keywords: Air Pollution (PM2.5); Atherosclerotic Surrogate; Brachial Flow-mediated Dilation; Carotid Intima-media Thickness; Montelukast Intervention; Atherosclerosis Prevention
MeSH Terms: conditions — Coronary Artery Disease | interventions — montelukast; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Montelukast (Active Comparator): Montelukast 10mg daily (tablet) orally x 26 weeks
  Interventions: Drug: Montelukast Oral Tablet
- Montelukast-matched placebo (Placebo Comparator): Placebo (Montelukast identical) tablet 1 daily orally x 26 weeks
  Interventions: Drug: Montelukast Placebo Oral Tablet

INTERVENTIONS:
Drug: Montelukast Oral Tablet — i) Montelukast 10mg daily (tablet) orally x 26 weeks
  Other Names: Montelukast (active)
  Arms: Montelukast
Drug: Montelukast Placebo Oral Tablet — i) Placebo (Montelukast identical) tablet 1 daily orally x 26weeks
  Other Names: Montelukast Placebo (control)
  Arms: Montelukast-matched placebo

SUMMARY:
Background: Longterm exposure to air pollution has been associated with cardiovascular events and mortality on top of traditional risk factors. Pulmonary inflammation and oxidative stress have been implicated. Brachial (arm) vascular reactivity (flow-mediated dilation FMD) and carotid (neck) artery intima-media thickness (CIMT) are highly reproducible atherosclerosis surrogates, predictive of cardiovascular and stroke outcome. Montelukast is proven safe and effective in alleviating pulmonary inflammation and oxidative stress when used in prevention of asthma episode.

Study objectives:

1. To test the hypothesis of pulmonary inflammation and oxidative stress-related vascular dysfunction in PM air pollution.
2. To evaluate the impact of Montelukast treatment as compared with placebo on predictive atherosclerosis surrogates (FMD and IMT).

Design: Parallel placebo control, randomized comparative study. Subjects will be randomized to take Montelukast (10mg/daily) or image-matched placebo for 26 weeks. Measures will include PM2.5/PM10, indices of subclinical atherosclerosis (brachial FMD and CIMT), blood inflammatory biomarkers (platelet counts, hsCRP and fibrinogen) and potential confounders (lipids and glucose).

Setting: 120 working adults aged 30-60 years in Hong Kong and 80 working adults in Chongqing (CREC Ref No: 2018.157, 2020.398)

Main outcome measures:

1. Subclinical atherosclerosis: (a) Endothelial function (brachial FMD) and (b) carotid intima media thickness (CIMT).
2. PM2.5 & PM10 concentrations: real-time measurement by portable devices twice at home and work sites.
3. Blood inflammatory markers-platelet count, hsCRP and Fibrinogen
4. Potential confounders: we shall collect informations on a range of potential confounders, including other air pollutants and traditional risk factors of atherosclerosis, entrusted to be controlled (stable).

Expected results: Adults after Montelukast treatment and exposed to high levels of PM2.5 or PM10 would have improved (increased) brachial FMD, and reduction of CIMT as compared with placebo. These will have great implication for comparative vascular epidemiology and development of preventive strategies.

DETAILED DESCRIPTION:
2. Introduction Atherosclerosis related complications, in particular stroke and coronary artery disease, are the most important health issues in modernized societies, being the leading cause of death worldwide. In addition to traditional cardiovascular (CV) risk factors such as obesity, hypertension, dyslipidemia, diabetes mellitus, tobacco use and physical inactivity, particulate matter (PM) air pollution has been shown to be associated with cardiovascular morbidity and mortality in large epidemiological studies.[1-3] Long-term exposure to elevated PM levels can reduce life expectancy, especially particulate matter with an aerodynamic diameter <2.5um (PM2.5). Such PM has a causal relationship to cardiovascular morbidity and mortality.[1-4] An approximate 8-18% increase in cardiovascular mortality has been observed for every 10ug/m3 elevation in average PM2.5 exposure over the long term. [1. 3, 5] The biological mechanisms of atherogenic processes may involve direct effects of PM on cardiovascular system, and/or indirect effects mediated by oxidative stress and inflammation. [6-7] Far less research has been conducted so far on the contribution of PM to such long-term atherogenic processes in human populations. [1,2,8,9]

We have previously studied 1656 Chinese adults in southern and northern China in 1996 to 2007 with PM2.5 concentration ranging from 34 to 94 ug/m3. PM2.5 were significantly related to prognostic atherosclerotic surrogates i.e. brachial flow-mediated dilatation (FMD) and carotid intima media thickness (IMT), independent of traditional-risk factors.[10] Our CATHAY study supports a hypothesis that PM2.5 air pollution is strongly correlated with early atherosclerotic process in modernizing China.

Montelukast has been used successfully and proven safe for prevention of asthma episodes, supposed to be triggered by allergic-related inflammations of respiratory tract. Similar inflammatory process at lung and subsequently at blood vessels may be implicated in PM2.5-related accelerated atherosclerosis. [9]

3. Aims and Hypotheses to be Tested: PM2.5 air pollution has been proven accelerating atherosclerotic process in Hong Kong and mainland China (CATHAY study). To further test this initial hypothesis, this interventional substudy aims

1) To evaluate the impact of antiinflammatory agent Montelukast treatment on predictive atherosclerosis surrogates (FMD & IMT).

2) To evaluate the mechanism involved in PM2.5-related vascular dysfunction by monitoring changes in systemic inflammatory markers (platelet counts, HsCRP and fibrinogen).

4. Plan of Investigation

4.1 The impact of interventional agents on FMD and carotid IMT in working adults Subjects (120 adults in Hong Kong and 80 adults in Chongqing)

Inclusion

* asymptomatic adults
* aged 30-60 years with
* gender: male or female
* concordance of home and workplace air pollution

High exposure group: 60 adults, with PM2.5 concentration exposure >30ug/m3, both at residence and at work.

Low exposure group: 60 sex and age-matched asymptomatic adults with PM2.5 exposure <30ug/m3 both at home and at work.

Exclusion:

* Those with family history of stroke, cardio-vascular disease
* Hypertension with blood pressure >150/90 mmHg
* Diabetes Mellitus
* Overweight/ obesity (BMI >25kg/M2)
* Cigarette smoking or ex-smoker <5 years
* Known dyslipidemia defined as LDL-C >4.1mmol/l and triglyceride >3.0mmol/l.
* Physical inactivity, with weekly leisure exercise less than 0.5 hour
* Continuous usage of vitamins or herbal medicines in recent one year.

Study design:

A flowchart figure in Annex 1 illustrates the major procedures for the proposed study. Brachial flow-mediated dilation before and after Montelukast intervention will be compared between the control and intervention group.

Methods After informed written consent, these participants (60 adults in Hong Kong, and 40 adults in Chongqing) will be randomized to take Montelukast 10mg/daily or image-matched placebo (60 adults in Hong Kong, and 40 adults in Chongqing) for 26 weeks.

Week-0 Week-13 Week-26 Health Examination + 0 + Vascular Study + 0 + Blood Test + 0 + PM2.5 Evaluation + 0 + Medicine Dispatch + + 0 Compliance Assessment 0 + +

* Collection of health data:

  1. Questionnaire - All adult subjects will be interviewed and required to complete a detailed questionnaire regarding their individual and family history of cardiovascular diseases, hypertension, diabetes and current use of medications. Information on socio-economic status and lifestyle will be collected. Important factors associated with PM exposure, such as transportation between work and home, environmental tobacco use (ETS), duration of residence, home renovation, cooking/heating usage, and use of incense and mosquito coils will be recorded as well.
  2. Health examination - Each participant will receive a health examination and their weight and height, blood pressures, body mass index (BMI) and wait-hip circumference ratio (WHR) will be measured when they are wearing light clothing and no shoes.
  3. Blood test: 10ml of fasting blood will be taken for platelet, fasting glucose, low density cholesterol, hsC-reactive protein and fibrinogen.
* Vascular Studies

  1. Endothelial function, (flow mediated dilation, FMD) of the brachial artery will be studied by using high resolution ultrasound, as described previously. [11, 12] Using a linear array transducer (L10-5) with a median frequency of 7.5MHz and a standard Advanced Technology Laboratories 3000 or Sonosite systems, and forearm tourniquet cuff placement to induce reactive hyperemia on deflation. Scans will be acquired at rest, during reactive hyperemia (to induce flow-mediated endothelium-dependent dilation, FMD). FMD will be expressed as % of dilation from baseline vessel diameter normalized with vessel strain.
  2. Carotid intima-media thickness (CIMT) measurement - B-mode ultrasound examinations will be performed using X12-3 probe with a 7 MHz scanning frequency linear array transducer. All carotid scans will be performed by standardized scanning protocol for the right and left carotid arteries as described by Salonen and Salonen [13] and Touboul et al [14], using images of the far wall of the distal 10 mm of the common carotid arteries, and a verified automatic edge-detecting and measurement software package as we described previously. [11-12, 15-16] The inter-observer variability of mean IMT is 0.003 to 0.011mm (CV 0.998%).
* Collection of air pollution exposure data:

Measurement of air pollutants at home and workplace will focus on PM2.5 and PM10.

We shall measure PM2.5 and PM10 pollutant levels at homes and workplace twice (warm and cool seasons) by handy portable PM2.5 device. The micro-environment meteorological PM2.5 and PM10 data, at home and workplace, will be combined and compared with data using modeling techniques.

Estimate of PM2.5/ PM10 exposure for each participant:

Details of the methodology and its verification using PM2.5/ PM10 data from Hong Kong and China has already been published (17, 18). Change of residential address during follow-up will be taken into account.

5. Significance and Potential: The proposed study can serve as a baseline for cohort model study in near future, for comparison with other vascular epidemiological data and interventional strategies in mainland China.

Investigating the relationship between particulate matter (PM) air pollution and atherosclerosis in working adulthood will enhance our abilities to elucidate the mechanisms underlying the effects of PM on atherosclerosis disease. Subsequently, it will help to develop appropriate strategies for both the control of PM air pollution (by legislation) and the prevention of atherosclerotic diseases, such as aerosol filters, facial masks, certain health food or nutrient (Aloe), statin or leukotriene modifiers (Montelukast) medicines. A huge number of Chinese exposed to PM air pollution throughout their life courses will be expected.

6. Compliance with Declaration of Helsinki The design, methodology and conduction of project are in compliance with Declaration of Helsinki.

7. Compliance will ICH-GCP. The medicines used are freely commercially available in Hong Kong Pharmacological Registry and compliant with ICH-GCP.

8. Data processing and analysis Power Calculation: The Proc Power in the STS 9.2 statistical packages (SAS institute Inc. Comy. NC, US) was used to calculate the sample size for FMD and carotid IMT. Data from our previous studies on adults in Hong Kong and mainland China, showed that the mean FMD is 6-8%+/-1.3% in otherwise healthy adults aged 30-60 years, and carotid IMT is 0.55-0.68mm+/-0.1mm. On the assumption of post Montelukast treatment, brachial FMD will improve to 6.7-8.7+/-1.4% in adults, and carotid IMT will reduce to 0.51-0.61mm+/-0.11mm, recruitment of 114 Chinese adults (57 in each group) will be adequately powered (80%) to detect a group difference in FMD of 1.2% and in CIMT of 0.1mm (12%) between the two treatment groups. In old adults, Kunzli reported a difference in CIMT of 12.1% in exposure of 20ug/m3 difference in PM2.5 pollution.[19]

Data Analysis: Statistical Analysis System 9.2 will be used for all statistical analyses. The primary endpoints are brachial FMD and Carotid IMT, serological inflammatory biomarkers (Platelet hsCRP and Fibrinogen) are secondary endpoints. Students' T-tests will be used to detect group differences on FMD and CIMT. Multivariate linear and logistic regression will be used to calculate risk magnitude by Montelukast vs placebo, and to control for potential confounders such as various traditional cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic Chinese adults
* aged 30-60 years with
* concordant ambient PM2.5 exposure, both at home and at workplace.

Exclusion Criteria:

* Those with family history of stroke, cardio-vascular disease
* Hypertension with blood pressure >150/90 mmHg
* Diabetics Mellitus
* Overweight/ obesity (BMI >25kg/M2)
* Cigarette smoking or ex-smoker <5 years
* Known dyslipidemia defined as fasting LDL-C >4.1mmol/l and triglyceride >3.0 mmol/l.
* Physical inactivity, with weekly leisure exercise less than 0.5 hour
* Continuous usage of vitamins or herbal medicines in recent one year

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Brachial flow-mediated dilation (FMD) | At baseline and 26 weeks of interventional treatment
  Changes in endothelial function (brachial FMD) in %
Carotid intima media thickness (CIMT) | At baseline and 26 weeks of interventional treatment
  Changes in carotid intima media thickness (CIMT) in mm

SECONDARY OUTCOMES:
Changes of platelet count in k/uL | At baseline and 26 weeks of interventional treatment
  Blood inflammatory markers
Changes of hsCRP in mg/ml | At baseline and 26 weeks of interventional treatment
  Blood inflammatory markers
Changes of Fibrinogen in g/l | At baseline and 26 weeks of interventional treatment
  Blood inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Kam Sang Woo, Principal Investigator — Adjunct Professor
Locations (1):
- The Chinese University of Hong Kong, Department of Medicine & Therapeutics, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: These materials will be available and shared on reasonable requests to Prof KS Woo from January 2024 till December 2024.
Access Criteria: These informations will be available and shared on reasonable requests to Prof KS Woo from January 2024 till December 2024. (kamsangwoo@cuhk.edu.hk/ crec@cuhk.edu.hk)

REFERENCES:
- [Result] Brook RD, Rajagopalan S, Pope CA 3rd, Brook JR, Bhatnagar A, Diez-Roux AV, Holguin F, Hong Y, Luepker RV, Mittleman MA, Peters A, Siscovick D, Smith SC Jr, Whitsel L, Kaufman JD; American Heart Association Council on Epidemiology and Prevention, Council on the Kidney in Cardiovascular Disease, and Council on Nutrition, Physical Activity and Metabolism. Particulate matter air pollution and cardiovascular disease: An update to the scientific statement from the American Heart Association. Circulation. 2010 Jun 1;121(21):2331-78. doi: 10.1161/CIR.0b013e3181dbece1. Epub 2010 May 10. PMID 20458016
- [Result] Rajagopalan S, Al-Kindi SG, Brook RD. Air Pollution and Cardiovascular Disease: JACC State-of-the-Art Review. J Am Coll Cardiol. 2018 Oct 23;72(17):2054-2070. doi: 10.1016/j.jacc.2018.07.099. PMID 30336830
- [Result] Franklin BA, Brook R, Arden Pope C 3rd. Air pollution and cardiovascular disease. Curr Probl Cardiol. 2015 May;40(5):207-38. doi: 10.1016/j.cpcardiol.2015.01.003. Epub 2015 Jan 3. PMID 25882781
- [Result] Pope CA 3rd, Burnett RT, Thurston GD, Thun MJ, Calle EE, Krewski D, Godleski JJ. Cardiovascular mortality and long-term exposure to particulate air pollution: epidemiological evidence of general pathophysiological pathways of disease. Circulation. 2004 Jan 6;109(1):71-7. doi: 10.1161/01.CIR.0000108927.80044.7F. Epub 2003 Dec 15. PMID 14676145
- [Result] Yu ITS, hui Zhang Y, San Tam WW, Yan QH, Xu YJ, Xun XJ, Wu W, Ma WJ, Tian LW, Tse LA, Lao XQ. Effect of ambient air pollution on daily mortality rates in Guangzhou, China. Atmos Environ 2012;46:528-535.
- [Result] Hajat A, Allison M, Diez-Roux AV, Jenny NS, Jorgensen NW, Szpiro AA, Vedal S, Kaufman JD. Long-term exposure to air pollution and markers of inflammation, coagulation, and endothelial activation: a repeat-measures analysis in the Multi-Ethnic Study of Atherosclerosis (MESA). Epidemiology. 2015 May;26(3):310-20. doi: 10.1097/EDE.0000000000000267. PMID 25710246
- [Result] Munzel T, Herzog J, Schmidt FP, Sorensen M. Environmental stressors and cardiovascular disease: the evidence is growing. Eur Heart J. 2017 Aug 1;38(29):2297-2299. doi: 10.1093/eurheartj/ehx306. No abstract available. PMID 28641401
- [Result] Pun VC, Yu IT, Ho KF, Qiu H, Sun Z, Tian L. Differential effects of source-specific particulate matter on emergency hospitalizations for ischemic heart disease in Hong Kong. Environ Health Perspect. 2014 Apr;122(4):391-6. doi: 10.1289/ehp.1307213. Epub 2014 Feb 7. PMID 24509062
- [Result] Kunzli N, Tager IB. Air pollution: from lung to heart. Swiss Med Wkly. 2005 Dec 10;135(47-48):697-702. doi: 10.4414/smw.2005.11025. PMID 16511705
- [Result] Woo KS, Chook P, Hu YJ, Lao XQ, Lin CQ, Lee P, Kwok C, Wei AN, Guo DS, Yin YH, Lau K, Leung KS, Leung Y, Celermajer DS. The impact of particulate matter air pollution (PM2.5) on atherosclerosis in modernizing China: a report from the CATHAY study. Int J Epidemiol. 2021 May 17;50(2):578-588. doi: 10.1093/ije/dyaa235. PMID 33349857
- [Result] Woo KS, Robinson JT, Chook P, Adams MR, Yip G, Mai ZJ, Lam CW, Sorensen KE, Deanfield JE, Celermajer DS. Differences in the effect of cigarette smoking on endothelial function in chinese and white adults. Ann Intern Med. 1997 Sep 1;127(5):372-5. doi: 10.7326/0003-4819-127-5-199709010-00006. PMID 9273828
- [Result] Woo KS, Chook P, Raitakari OT, McQuillan B, Feng JZ, Celermajer DS. Westernization of Chinese adults and increased subclinical atherosclerosis. Arterioscler Thromb Vasc Biol. 1999 Oct;19(10):2487-93. doi: 10.1161/01.atv.19.10.2487. PMID 10521379
- [Result] Salonen JT, Salonen R. Ultrasonographically assessed carotid morphology and the risk of coronary heart disease. Arterioscler Thromb. 1991 Sep-Oct;11(5):1245-9. doi: 10.1161/01.atv.11.5.1245. PMID 1911709
- [Result] Touboul PJ, Hennerici MG, Meairs S, Adams H, Amarenco P, Desvarieux M, Ebrahim S, Fatar M, Hernandez Hernandez R, Kownator S, Prati P, Rundek T, Taylor A, Bornstein N, Csiba L, Vicaut E, Woo KS, Zannad F; Advisory Board of the 3rd Watching the Risk Symposium 2004, 13th European Stroke Conference. Mannheim intima-media thickness consensus. Cerebrovasc Dis. 2004;18(4):346-9. doi: 10.1159/000081812. Epub 2004 Nov 2. PMID 15523176
- [Result] Thomas GN, Chook P, Qiao M, Huang XS, Leong HC, Celermajer DS, Woo KS. Deleterious impact of "high normal" glucose levels and other metabolic syndrome components on arterial endothelial function and intima-media thickness in apparently healthy Chinese subjects: the CATHAY study. Arterioscler Thromb Vasc Biol. 2004 Apr;24(4):739-43. doi: 10.1161/01.ATV.0000118015.26978.07. Epub 2004 Jan 22. PMID 14739120
- [Result] Woo KS, Chook P, Yu CW, Sung RY, Qiao M, Leung SS, Lam CW, Metreweli C, Celermajer DS. Effects of diet and exercise on obesity-related vascular dysfunction in children. Circulation. 2004 Apr 27;109(16):1981-6. doi: 10.1161/01.CIR.0000126599.47470.BE. Epub 2004 Apr 5. PMID 15066949
- [Result] [17] Lin CQ, Li Y, Yuan ZB, Lau AKH, Li, CC, and Fung JCH. Using satellite remote sensing data to estimate the high-resolution distribution of ground-level PM2.5. Remote Sens. Environ 2015;156:117-128.
- [Result] [18] Lin CQ, Liu G, Lau AKH, Li Y, Li CC, Fung JCH, and Lao XQ. High-resolution satellite remote sensing of provincial PM2.5 trends in China from 2001 to 2015. Atmos. Environ 2018;180:110-116
- [Result] Kunzli N, Jerrett M, Mack WJ, Beckerman B, LaBree L, Gilliland F, Thomas D, Peters J, Hodis HN. Ambient air pollution and atherosclerosis in Los Angeles. Environ Health Perspect. 2005 Feb;113(2):201-6. doi: 10.1289/ehp.7523. PMID 15687058